CLINICAL TRIAL: NCT05873075
Title: The Effects of Intravascular Laser Irradiation of Blood on Reproductive Outcomes in Poor Ovaria n Responders Undergoing in Vitro Fertilization Cycles
Brief Title: Intravascular Laser Irradiation of Blood Use in Poor Ovarian Responders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Principal Investigator, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH23-CT3-20
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Unrecognized Condition
Keywords: Intravascular laser irradiation of blood; He-Ne laser; Poor ovarian responder; Assisted reproductive technology; In vitro fertilization; Anti-aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients received intravascular laser irradiation of blood for 20 days before IVF cycles
  Interventions: Other: Intravascular laser irradiation of blood
- Control (No Intervention): No intervention before IVF cycles

INTERVENTIONS:
Other: Intravascular laser irradiation of blood — Intravascular laser irradiation of blood via an intravenous catheter for irradiation of the blood under a period of 60 minutes daily for 20 days
  Arms: Study group

SUMMARY:
The aim of this study was to investigate the effects of intravascular laser irradiation of blood on outcomes of in vitro fertilization cycles in poor ovarian responders.

DETAILED DESCRIPTION:
Intravascular laser irradiation of blood (ILIB) with He-Ne laser (632.8nm) has been applied on many organs and on the hematologic and immunologic system. Quite a number of both animal and human experiments have demonstrated that ILIB has a wide range of effects, including biostimulation, analgesia, antiallergic effects, immunomodulation, vasodilatation, antihypoxic, anti-oxidant, anti-aging and anti-inflammatory effects.

Poor ovarian responders (PORs) defined as poor or no response to ovarian stimulation had poor prognosis in assisted artificial technique (ART), which is a great challenge in in vitro fertilization (IVF) cycles. Previous studies showed that treatment with anti-oxidants could improve the outcomes of the poor ovarian responders; however, the effect is limited. Since ILIB has anti-aging, anti-oxidant and anti-inflammatory effects, the investigators hypothesize that ILIB may improve ovarian function and oocyte quality in PORs. Therefore, the investigators attempt to explore the effects of ILIB on the IVF outcomes in women with poor ovarian response.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergoes IVF cycles
* BMI:18-30 kg/m2
* Diminished ovarian reserve (AFC<5, AMH<1.2 ng/ml)

Exclusion Criteria:

* Primary ovarian insufficiency
* Congenital uterine anomaly
* Severe intrauterine adhesion
* Severe male factor (azoospermia)
* Chromosome anomaly
* Malignancy
* Donor cycles

Ages: 30 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | through study completion, an average of 1 year
  continuous presence of a fetal heartbeat over 12 weeks of a pregnancy
Ovarian reserve marker | through study completion, an average of 1 year
  Anti-mullerian hormone levels

SECONDARY OUTCOMES:
mitochondrial function of cumulus cells | through study completion, an average of 1 year
  Oxygen consumption and adenosine triphosphate production

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Momenzadeh S, Abbasi M, Ebadifar A, Aryani M, Bayrami J, Nematollahi F. The intravenous laser blood irradiation in chronic pain and fibromyalgia. J Lasers Med Sci. 2015 Winter;6(1):6-9. PMID 25699161
- [Background] Mikhaylov VA. The use of Intravenous Laser Blood Irradiation (ILBI) at 630-640 nm to prevent vascular diseases and to increase life expectancy. Laser Ther. 2015 Mar 31;24(1):15-26. doi: 10.5978/islsm.15-OR-02. PMID 25941421
- [Background] Huang SF, Tsai YA, Wu SB, Wei YH, Tsai PY, Chuang TY. Effects of intravascular laser irradiation of blood in mitochondria dysfunction and oxidative stress in adults with chronic spinal cord injury. Photomed Laser Surg. 2012 Oct;30(10):579-86. doi: 10.1089/pho.2012.3228. Epub 2012 Aug 14. PMID 22891782
- [Background] Tsai HW, Wang PH, Hsu PT, Chen SN, Lin LT, Li CJ, Tsui KH. Laser irradiation pretreatment improves endometrial preparation of frozen-thawed embryo transfer in recurrent implantation failure patients. Gynecol Endocrinol. 2020 Aug;36(8):734-738. doi: 10.1080/09513590.2020.1712694. Epub 2020 Jan 13. PMID 31928249